CLINICAL TRIAL: NCT06160505
Title: Mastoidectomy Followed by Mastoid Obliteration Using S53P4 Bioactive Glass Versus Mastoidectomy Alone for Chronic Suppurative Otitis Media: a Retrospective Comparative Study
Brief Title: Mastoid Obliteration Using S53P4 Bioactive Glass Versus Mastoidectomy Alone for Chronic Suppurative Otitis Media
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diakonessenhuis, Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: 16-004-2
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Chronic Suppurative Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients that underwent mastoidectomy alone: This is the control group, consisting of patients that have underwent either canal wall up or canal wall down mastoidectomy for CSOM without mastoid obliteration
- Patients that underwent mastoidectomy + mastoid obliteration: This is the intervention group, consisting of patients that have underwent either canal wall up or canal wall down mastoidectomy for CSOM followed by obliteration of the mastoid cavity using S53P4 bioactive glass
  Interventions: Device: S53P4 Bioactive glass

INTERVENTIONS:
Device: S53P4 Bioactive glass — Following mastoidectomy, the mastoid cavity, and if the ossicular chain has been removed the epitympanum as well, are obliterated using S53P4 bioactive glass. The bioactive glass is mixed with saline and administered to the cavity, ensuring a tight fit.
  Groups: Patients that underwent mastoidectomy + mastoid obliteration

SUMMARY:
Chronic suppurative otitis media (CSOM) is characterized by intermittent or continuous otorrhea lasting for longer than 6 weeks. Most cases can be treated conservatively using antibiotic drops and oral antibiotics. However, some cases will not respond to conservative treatment and demonstrate persistant discharge. In these cases, especially if a CT-scan shows opacification of the mastoid air cells, a mastoidectomy can be considered as treatment modality. In recent years, obliteration of the mastoid cavity following mastoidectomy is gaining popularity. However, the effectiveness of obliterating the mastoid in comparison to mastoidectomy alone is uncertain for CSOM. In this retrospective cohort study, our aim is to compare mastoidectomy to mastoidectomy + mastoid obliteration in a cohort of patients suffering from CSOM with mastoid involvement. The hypothesis is that obliterating the mastoid cavity will result in a higher frequency of dry ears and in a lower frequency of revision surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from CSOM, as indicated by otorrhea as main complaint preoperatively
* At least one year of follow-up, in order to asses the primary outcome
* Opacification of the mastoid air cells on preoperative CT-scans, as indication for mastoid involvement
* Canal wall up or canal wall down mastoidectomy
* Operated between 2010 and 2022

Exclusion Criteria:

* Patients suffering from middle ear cholesteatoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent canal wall up or canal wall down mastoidectomy between 2010 and 2022 will be evaluated. Only cases that full-fill the in- and exclusion criteria will be selected. Patients will be stratified for whether they received mastoid obliteration or not.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with a dry ear at one-year postoperatively | At 1-year postoperatively
  The number of cases that have a dry ear at the one-year postoperative out-patient visit. A dry ear is defined as Merchant grade 0 or 1 (No otorrhea or less than one period of otorrhea in the last three months, respectively). A wet ear, thus suffering from otorrhea, is defined as merchant grade 2 or 3 (intermittent more than once in last three months or continuous discharge, respectively). We compare the obliteration cohort to the non-obliteration cohort.

SECONDARY OUTCOMES:
The number of cases with perforations of the tympanic membrane during follow-up | Measured at 1-year postoperatively and 3-years postoperatively
  The number of cases that will develop a perforation of the tympanic membrane during follow-up
  We compare the obliteration cohort to the non-obliteration cohort.
The difference in air conduction postoperatively | First audiometry postoperatively, which is made at 6 months postoperatively
  The differences in air conduction postoperatively, as measured in the first audiometry postoperatively in decibel.
  We compare the obliteration cohort to the non-obliteration cohort.
The number of cases which require revision surgery during follow-up | Measured at 3-years and 5-years postoperatively
  The number of cases which require revision surgery during follow-up, for either recurrent CSOM and other indications
  We compare the obliteration cohort to the non-obliteration cohort.

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Quak, MD, PhD, Principal Investigator — Diakonessenhuis, Utrecht
Locations (1):
- Diakonessenhuis, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided